CLINICAL TRIAL: NCT06628128
Title: An Open-Label Extension Study to Evaluate the Long-Term Safety and Efficacy of JNT-517 in Participants With Phenylketonuria
Brief Title: A Study to Evaluate the Long-Term Safety and Efficacy of JNT-517 in Participants With Phenylketonuria
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JNT517-501
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Phenylketonuria (PKU)
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Adult: 75 mg BID (Experimental)
  Interventions: Drug: JNT-517 Tablet
- Adult: 150 mg BID (Experimental)
  Interventions: Drug: JNT-517 Tablet
- Adolescent: 75 mg BID (Experimental)
  Interventions: Drug: JNT-517 Tablet
- Adolescent: 150 mg BID (Experimental)
  Interventions: Drug: JNT-517 Tablet

INTERVENTIONS:
Drug: JNT-517 Tablet — JNT-517: 75 mg BID

SUMMARY:
The goal of this Phase 3, open-label extension study is to evaluate the long-term safety and efficacy of JNT-517 in participants with Phenylketonuria (PKU) after completion of either Study JNT517-101 or JNT517-201. In this long-term extension (LTE) study, all adults (aged ≥18 years) who complete Study JNT517-101 will be randomized 1:1 to receive JNT-517 at 75 mg twice daily (BID) or 150 mg BID, regardless of their previous dose. Adolescent participants who complete Study JNT517-201 will receive the same JNT-517 dose of the cohort they were initially assigned to, either 75 mg BID or 150 mg BID.

ELIGIBILITY:
Key Inclusion Criteria:

1. Clinical diagnosis of PKU and has completed Study JNT517-101 or Study JNT517-201.
2. Not on pegvaliase within 4 weeks of Screening.
3. If on sapropterin or large neutral amino acids at Screening, must be on a stable dose for 4 weeks prior to Screening and expected to be on stable dose for the study duration.
4. Willing and able to maintain a diet consistent in protein content from natural intact and medical food protein sources from the Screening period through the duration of the study under the direction of a dietician.
5. If female of childbearing potential:

   1. Must have a negative serum pregnancy test at Screening and a negative urine pregnancy test by Day 1.
   2. Must practice sexual abstinence, or if involved in any sexual intercourse that could lead to pregnancy, must agree to use 2 highly effective contraceptive methods (see Section 7.3.1 for details of contraception) from Screening until at least 30 days after the last study drug administration.
   3. If taking estrogen- or progesterone-based oral contraceptives, must agree to use 2 other highly effective methods of contraception or must agree to sexual abstinence during the study.
6. Is a female not of childbearing potential or postmenopausal, defined as follows:

   1. Has had surgical sterilization (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy).
   2. Has had amenorrhea for minimum of 1 year with confirmation by levels of follicle stimulating hormone testing.
   3. Has not achieved menarche (has not had first menstrual period). If a female achieves menarche during the study, she will need to follow the contraception requirement for females of childbearing potential.
7. If male, must practice sexual abstinence, or if involved in any sexual intercourse that could lead to pregnancy, must agree to use highly effective contraceptive methods from Day 1 until at least 30 days after the last study drug administration.

   Note: No restrictions are required for males who have undergone a documented vasectomy at least 4 months prior to Screening. If the vasectomy procedure is not documented or was performed less than 4 months prior to Screening, males must follow the same contraception as for non-vasectomized participants.
8. Capable of giving signed informed consent or and/or assent (for adolescents) and able to comply with study procedures.
9. Participants with psychiatric illness must be well-controlled for the last 3 months prior to screening visit and if on medication, on stable medications for the last 3 months.

Key Exclusion Criteria:

1. Continuation into the LTE is not considered safe and/or feasible in the opinion of the Investigator.
2. Any acute or chronic medical condition that would prevent the participant from complying with the procedures or place the participant at risk if they participate in the study.
3. Positive for hepatitis B or C or human immunodeficiency virus.
4. Any history of liver disease.
5. Any history of cataracts or more than minimal cataracts observed during the Screening ophthalmologic examination. Minimal cataracts are defined as changes similar to LOCS II (lens opacities classification system II) lens grade C1, N1, or P1, or an equivalent grading system.
6. Any surgical or medical conditions that may affect study drug absorption, distribution, metabolism, or excretion.
7. Creatinine clearance ˂90 mL/min by 2021 Chronic Kidney Disease Epidemiology Collaboration formula for adults and by the Schwartz formula for adolescents (˂18 years of age)
8. History of drug or alcohol abuse in the last year.
9. Use of any medication that are inhibitors or inducers of cytochrome P450 (CYP)3A4 or inhibitors of the transporter P glycoprotein (P-gp) within 4 weeks prior to randomization and unwilling and/or unable to avoid these medications throughout the treatment duration.
10. Use of any medication that is a substrate of CYP3A4, or a substrate of the transporters P gp, breast cancer resistance protein (BCRP), organic anion transporter 3 (OAT3), multidrug and toxin extrusion (MATE)1, or MATE2-K within 4 weeks prior to randomization and unwilling and/or unable to avoid these medications throughout the treatment duration.
11. Current, recent, or suspected infection within 2 weeks of Screening of SARS-CoV-2/COVID-19.
12. Unable to tolerate oral medication or inability to swallow tablets.
13. Allergy to JNT-517 or any component of the investigational product.
14. Any of the following laboratory values at the Screening visit:

    1. Alanine aminotransferase or aspartate aminotransferase values ˃ the upper limit of normal (ULN)
    2. Total bilirubin ˃ULN
    3. Hemoglobin ˂11.0 g/dL (˂110.0 g/L)
    4. White blood cell count ˃ULN
    5. Platelet count ˂150 × 109/L (˂150,000/mm3)
15. Participation in another investigational drug trial within 30 days (other than for JNT-517) or, if known 5 half-lives of investigational drug (whichever is longer).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Screening to +2 weeks from last dose
  Reported based on results of 12-lead electrocardiograms (ECGs), vital signs, clinical laboratory tests, and other medical assessments.

SECONDARY OUTCOMES:
Change from baseline in plasma Phe and other amino acids | Baseline to +2 weeks from last dose
Change from baseline in urinary Phe and other amino acids | Baseline to +2 weeks from last dose
Change from baseline in dietary Phe and protein intake | Baseline to +2 weeks from last dose

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on the Vivli data sharing platform which can be found here: https://vivli.org/ourmember/Otsuka/
URL: http://clinical-trials.otsuka.com